CLINICAL TRIAL: NCT03992560
Title: A Prospective Randomised Multi-centre Trial Comparing cArdiac MRI Guided CRT Versus Conventional CRT Implantation in Patients With Ischaemic Cardiomyopathy
Acronym: TACTIC CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.1
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard CRT implantation (No Intervention)
- MRI guided CRT implantation (Experimental)
  Interventions: Device: Guide CRT Software Prototype

INTERVENTIONS:
Device: Guide CRT Software Prototype — The medical device in the trial is a software programme that allows image fusion of previously acquired MRI images with real-time X-Ray fluoroscopic images in the cardiac catheter laboratory. We are able to use the MRI information to assess the best location to place the left ventricular lead for a CRT device and then superimpose this location onto the real-time X-Ray fluoroscopic images during the left ventricular lead implantation
  Arms: MRI guided CRT implantation

SUMMARY:
The purpose of the study is to determine whether MRI guided CRT implantation (using Siemen's software prototype) is superior to standard treatment in terms of CRT response. Data will be collected at enrolment, implant, pre-discharge, 6 weeks and 6 months. The total duration of the investigation will be 6 months.

The primary endpoint will be assessed by calculating the difference in the proportion of responders (>15% reduction in end systolic volume derived from 2-dimensional transthoracic echocardiogram at 6 months post CRT implant).

ELIGIBILITY:
Inclusion Criteria:

* >18yrs of age
* Standard indication for CRT-P or CRT-D according to European Society of Cardiology (ESC)/European Heart Rhythm (EHRA) guidelines.1
* Stable on optimal medical therapy for at least 3 months
* Ischaemic aetiology
* Patients with atrial fibrillation can be included

Exclusion Criteria:

* Any contraindication to pacing /implantable cardioverter-defibrillator (ICD) implant
* Requirement for endocardial pacing
* Contraindication to gadolinium contrast enhanced cardiac Magnetic Resonance (MR) scanning
* Significant claustrophobia
* Significant renal impairment with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2
* Existing pacemaker or ICD system or extraction of a CRT system within the last 6 months
* Participation in other studies with active treatment/ investigational arm
* Pregnant or planning to become pregnant in the next 7 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2024-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
>15% reduction in end systolic volume | 6 months
  >15% reduction in end systolic volume derived from 2-dimensional transthoracic echocardiogram at 6 months post CRT implant

SECONDARY OUTCOMES:
5% absolute increase in left ventricular ejection fraction | 6 months
  5% absolute increase in left ventricular ejection fraction as derived from 2D echocardiogram
>10% reduction in end diastolic volume | 6 months
  >10% reduction in end diastolic volume as derived from 2D echocardiogram

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No